CLINICAL TRIAL: NCT04425057
Title: Effect of a High Intensity Interval Training in Older Adults With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, PhD, PT, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/0113
Record Dates: First submitted 2018-12-31; First posted 2020-06-11 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval training (Experimental): Physiotherapy program during two months: Interval training at a high intensity, inlcuding a warm-up and a cool-down. Aerobic exercises, resistance exercises, stretching
  Interventions: Other: Interval training
- Control group (No Intervention): No physiotherapy

INTERVENTIONS:
Other: Interval training
  Arms: Interval training

SUMMARY:
A study comparing 2 groups: interval training and control group. Interval training group will perform a physiotherapy program based in exercises, at a high intensity, and stretching of muscles at the end. Control group will not perform any physiotherapy program. Several parameters will be evaluated at baseline, 2 months and 6 months: anxiety, depression, functional capacity, blood pressure, lipid profile, physical activity, ecc.

DETAILED DESCRIPTION:
A study comparing 2 groups: high intensity interval training and control group. Interval training group will perform a two-month physiotherapy program based in exercises, at a high intensity, and stretching of muscles at the end. Intensity will be established based on Borg scale and an effort test.

Control group will not perform any physiotherapy program, but will have usual care with medication.

Several parameters will be evaluated at baseline, 2 months and 6 months: anxiety, depression, functional capacity, blood pressure, lipid profile, physical activity, ecc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of coronary artery disease
* Discharged from hospital, less than 2 months

Exclusion Criteria:

* Not able to move by themselves

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | baseline
  Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Kinesiophobia | 2 months
  Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Kinesiophobia | 6 months
  Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
body mass index | baseline
  body mass index, m/kg2
body mass index | 2 months
  body mass index, m/kg2
body mass index | 6 months
  body mass index, m/kg2
abdominal circumference | baseline
  abdominal circumference in cm
abdominal circumference | 2 months
  abdominal circumference in cm
abdominal circumference | 6 months
  abdominal circumference in cm
body fat | baseline
  Bioimpedanciometer OMRON HBF-500INT body fat in %
body fat | 2 months
  Bioimpedanciometer OMRON HBF-500INT body fat in %
body fat | 6 months
  Bioimpedanciometer OMRON HBF-500INT body fat in %
visceral fat | baseline
  Bioimpedanciometer OMRON HBF-500INT visceral fat in %
visceral fat | 2 months
  Bioimpedanciometer OMRON HBF-500INT visceral fat in %
visceral fat | 6 months
  Bioimpedanciometer OMRON HBF-500INT visceral fat in %
muscle mass | baseline
  Bioimpedanciometer OMRON HBF-500INT muscle mass in %
muscle mass | 2 months
  Bioimpedanciometer OMRON HBF-500INT muscle mass in %
muscle mass | 6 months
  Bioimpedanciometer OMRON HBF-500INT muscle mass in %

SECONDARY OUTCOMES:
anxiety | baseline
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
anxiety | 2 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
anxiety | 6 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
depression | baseline
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
depression | 2 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
depression | 6 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
physical activity | baseline
  International physical activity questionnaire: it has 9 items and provides information on the time spent while walking, in activities of low, moderate and vigorous intensity and in sedentary activities. Based on the estimated METS consumed, the IPAQ divides the subjects into three levels or categories: Low, moderate and high physical activity. The score of the different types of activity is expressed in METS-minutes per week.
physical activity | 2 months
  International physical activity questionnaire: it has 9 items and provides information on the time spent while walking, in activities of low, moderate and vigorous intensity and in sedentary activities. Based on the estimated METS consumed, the IPAQ divides the subjects into three levels or categories: Low, moderate and high physical activity. The score of the different types of activity is expressed in METS-minutes per week.
physical activity | 6 months
  International physical activity questionnaire: it has 9 items and provides information on the time spent while walking, in activities of low, moderate and vigorous intensity and in sedentary activities. Based on the estimated METS consumed, the IPAQ divides the subjects into three levels or categories: Low, moderate and high physical activity. The score of the different types of activity is expressed in METS-minutes per week.
functional capacity | baseline
  Incremental shuttle walk test will be used to measure functional capacity. Patients were required to walk along a level 10 m course at a previously determined speed dictated by signals from an audio tape recorder. The walking speed was progressively increased at 1 min intervals, for a total of 12 stages. The test was terminated if the patient was unable to continue at the desired speed or if the patient failed to complete the shuttle course in the allowed time.
  Distance walked were determined on exercise cessation (meters).
functional capacity | 2 months
  Incremental shuttle walk test will be used to measure functional capacity. Patients were required to walk along a level 10 m course at a previously determined speed dictated by signals from an audio tape recorder. The walking speed was progressively increased at 1 min intervals, for a total of 12 stages. The test was terminated if the patient was unable to continue at the desired speed or if the patient failed to complete the shuttle course in the allowed time.
  Distance walked were determined on exercise cessation (meters).
functional capacity | 6 months
  Incremental shuttle walk test will be used to measure functional capacity. Patients were required to walk along a level 10 m course at a previously determined speed dictated by signals from an audio tape recorder. The walking speed was progressively increased at 1 min intervals, for a total of 12 stages. The test was terminated if the patient was unable to continue at the desired speed or if the patient failed to complete the shuttle course in the allowed time.
  Distance walked were determined on exercise cessation (meters).
brachial systolic and diastolic blood pressure | baseline
  systolic and diastolic blood pressure (mmHg)
brachial systolic and diastolic blood pressure | 2 months
  systolic and diastolic blood pressure (mmHg)
brachial systolic and diastolic blood pressure | 6 months
  systolic and diastolic blood pressure (mmHg)
health related quality of life | baseline
  Short-form 36: the questionnaire is composed of 36 questions that value both positive and negative health status. It was developed from an extensive battery of questionnaires employed at WHO, which included 40 concepts related to health. The questionnaire contains 8 scales, which represent the concepts of health most frequently used in the main health questionnaires. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role, Mental health. The scores of each of the 8 dimensions of the SF-36 oscillate between 0 and 100. A result of 100 indicates optimal health and 0 would reflect a very poor state of health.
health related quality of life | 2 months
  Short-form 36: the questionnaire is composed of 36 questions that value both positive and negative health status. It was developed from an extensive battery of questionnaires employed at WHO, which included 40 concepts related to health. The questionnaire contains 8 scales, which represent the concepts of health most frequently used in the main health questionnaires. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role, Mental health. The scores of each of the 8 dimensions of the SF-36 oscillate between 0 and 100. A result of 100 indicates optimal health and 0 would reflect a very poor state of health.
health related quality of life | 6 months
  Short-form 36: the questionnaire is composed of 36 questions that value both positive and negative health status. It was developed from an extensive battery of questionnaires employed at WHO, which included 40 concepts related to health. The questionnaire contains 8 scales, which represent the concepts of health most frequently used in the main health questionnaires. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role, Mental health. The scores of each of the 8 dimensions of the SF-36 oscillate between 0 and 100. A result of 100 indicates optimal health and 0 would reflect a very poor state of health.

IPD SHARING:
Plan to Share IPD: No